CLINICAL TRIAL: NCT06676046
Title: Natural History of Uncommon Dyslipidemias, Rare Lipid Disorders and Unusual Atherosclerotic Conditions
Status: Recruiting | Type: Observational
Sponsor: National Heart, Lung, and Blood Institute (NHLBI) (NIH)
Responsible Party: Sponsor
Organization: National Institutes of Health Clinical Center (CC) (NIH)
Other Study IDs: 10001933; 001933-H
Record Dates: First submitted 2024-11-05; First posted 2024-11-06 (Actual); Last update posted 2025-08-01 (Actual); Status verified 2025-07-18

CONDITIONS: Dyslipidemia; Atherosclerosis
Keywords: Uncommon Dyslipidemias; Rare Lipid Disorders; Unusual Atherosclerotic Conditions; Lipoproteins; Atherosclerosis; TRIGLYCERIDES
MeSH Terms: conditions — Dyslipidemias; Atherosclerosis

STUDY DESIGN:
Observational Model: Other | Time Perspective: Prospective
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Patients diagnosed with rare primary lipid disorders.: Male and female participants with rare primary lipid disorders ages 10 and older.

SUMMARY:
Background:

The right amount of fats in the blood (cholesterol and triglycerides) are a key part of a healthy organism. Too much or too little of these fats may manifest as diseases (dyslipidemia). There are many causes for these abnormalities, but some are genetically determined and we would like to better understand the progression of these conditions over time.

Objective:

This natural history study aims to learn more about dyslipidemias; how they change over time; and how they respond to therapy. We also want to develop new diagnosis methods for these conditions. With the knowledge we will acquire we hope to provide new insights, new approaches and improve the overall health of these patients.

Eligibility:

Individuals aged 10 years and older, residing both within and outside the United States, who have or are suspected of having a disorder that causes changes in the levels of fats in their blood (genetic dyslipidemias).

Design:

Participants residing within and outside the United States will be screened. Their medical records may be reviewed. They may talk to researchers about their medical history by phone, telehealth, or in person.

All study visits are optional. Participants may visit the NIH up to 15 times per year, if needed.

Each visit may include a physical exam and blood tests. Participants may also have an electrocardiogram (EKG). The EKG measures the electrical activity when the heart beats.

In some cases, participants may remain in the study for up to 20 years.

DETAILED DESCRIPTION:
Study Description:

This clinical research project is designed as a rare primary lipid disorder patient observational study that will utilize conventional and virtual (TeleHealth) medicine. This study will accept patients from the U.S. and abroad, will utilize current approved regulatory approaches to receive patient data, specimens, and share information with patients or their healthcare providers.

Objectives:

-Primary objective:

To improve understanding of rare or uncommon or acquired primary lipid disorders, evolution of such conditions, and response to therapies among the participants enrolled onto this study based upon LDL-C and other lipids or lipoproteins over time.

-Secondary objective:

To improve understanding of how HDL-C, triglycerides, other lipid markers of dyslipidemia, and cardiovascular (CV) risk impact rare or uncommon or acquired primary lipid disorders, and response to therapies over time.

-Tertiary/Exploratory objectives:

Changes in nuclear magnetic resonance spectroscopy lipoprotein fractioning parameters, genetic markers, efflux rate, and other parameters related with CV risk.

* To study lipid and cardiovascular risk markers throughout pregnancy
* To develop new assays and screening tools for these rare, unusual and uncommon conditions.

Endpoints:

* Primary endpoints: Observe the changes in LDL-C overtime
* Secondary endpoints: Observe the changes in HDL-C, triglycerides, and other lipid markers of dyslipidemia and CV risk.
* Tertiary/Exploratory endpoints:

Observe changes in LDL-p, LDL-z, HDL-p, HDL-z, ApoA-I levels, ApoB levels, efflux rate. Observe known genetic markers associated with rare lipid disorders. Develop new assays or screening tools.

Observe changes in LDL-p, LDL-z, HDL-p, HDL-z, ApoA-I levels, ApoB levels, efflux rate, hs-CRP during pregnancy

ELIGIBILITY:
* INCLUSION CRITERIA:

Affected Participants

* Male and female participants age >= 10 years.
* Subjects with confirmed or suspected rare disorder that causes lipid/lipoprotein abnormalities (dyslipidemia) or abnormal documented or referred atherosclerosis patterns.
* Only affected individuals (not healthy volunteers and for self-referred subjects independent of lipid and lipoprotein marker values.); subjects with laboratory or clinical presentation that in the opinion of the Principal Investigator, would alter the determination of normal

parameters for assays and screening tools development.

-Ability of the subject or Legally Authorized Representative (LAR) to understand and willingness to sign a written informed consent document.

Healthy Volunteers

* Participants must be healthy, with no known history of lipid disorders or related medical conditions.
* Participants must not be pregnant.

EXCLUSION CRITERIA:

* Patients with disorders that cause common secondary/lipoprotein alterations.
* Patients with any other findings that, in the opinion of the Principal Investigator, would preclude them from participating in the study.

Ages: 10 Years to 90 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: Individuals with rare and/or unusual lipid disorders residing both within and outside the United States
Sampling Method: Non-Probability Sample
Enrollment: 1500 (Estimated)
Dates: Start 2025-01-15 (Actual); Primary Completion 2044-11-24 (Estimated); Study Completion 2044-11-24 (Estimated)

PRIMARY OUTCOMES:
Change overtime in low-density lipoprotein cholesterol (LDL-C). | up to 20 years
  To observe change overtime in low-density lipoprotein cholesterol (LDL-C).

SECONDARY OUTCOMES:
Change overtime in high-density lipoprotein cholesterol (HDL-C) | up to 20 years
  To observe the changes overtime in in high-density lipoprotein cholesterol (HDL-C)
Change overtime in triglycerides | up to 20 years
  To observe the changes overtime in triglycerides
Change overtime in lipid markers of dyslipidemia and cardiovascular risk. | up to 20 years
  To observe the changes overtime in lipid markers of dyslipidemia and cardiovascular risk.

CONTACTS AND LOCATIONS:
Overall Officials: Marcelo J Amar, M.D., Principal Investigator — National Heart, Lung, and Blood Institute (NHLBI)
Locations (1):
- National Institutes of Health Clinical Center, Bethesda, Maryland, United States

IPD SHARING:
Plan to Share IPD: Yes
All individual participant data (IPD) that underpin the results presented in a publication will be made available.
Supporting Information: Study Protocol, SAP, ICF
Time Frame: Starting approximately 6 months after publication and available indefinitely.
Access Criteria: Data will be shared through NHLBI BioData Catalyst, which is a controlled access repository.

REFERENCES:
- See also: NIH Clinical Center Detailed Web Page — https://clinicalstudies.info.nih.gov/cgi/detail.cgi?A_001933-H.html